CLINICAL TRIAL: NCT02655458
Title: Phase 1 Study of Elotuzumab in Combination With Autologous Stem Cell Transplantation and Lenalidomide Maintenance for Multiple Myeloma
Brief Title: Elotuzumab in Autologous Stem Cell Transplantation (ASCT) and Lenalidomide Maintenance for Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hearn Jay Cho (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Hearn Jay Cho, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-1275
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Induction Therapy; Autologous Stem Cell Transplant; ASCT; Auto-SCT
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous PBMC reconstitution, Elotuzumab, Lenalidomide (Experimental): Max number of cycles is 12. Elotuzumab will be administered IV 20 mg/kg on Day 1 of each cycle. Lenalidomide dosing will start with cycle 4 at 10 mg orally daily days 1-21.
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide; Other: autologous PBMC reconstitution; Other: ASCT

INTERVENTIONS:
Drug: Elotuzumab — The following must also be administered before any elotuzumab:
  Dexamethasone 8 mg IV (on the day of elotuzumab infusion 45-90 mins prior to the start of infusion), the following 30 - 90 minutes prior to start of infusion: H1 blocker: diphenhydramine (25 - 50 mg po or IV) or equivalent, H2 blocker: ranitidine (50 mg IV) or equivalent (adjusted for renal failure as indicated), acetaminophen (650 - 1000 mg po).
  Other Names: Empliciti
Drug: Lenalidomide — On the days of elotuzumab administration, the dose of lenalidomide is to be administered at least 2 hours after completion of elotuzumab dosing. Aspirin 81 mg PO daily will also be prescribed for DVT prophylaxis.
  Other Names: Revlimid
Other: autologous PBMC reconstitution — Autologous peripheral blood mononuclear cell collection and reconstitution. PBMC will be collected from patients by standard apheresis procedures. Up to 25 ml of autologous plasma will also be recovered for dilution of cryopreserved products (if necessary). For reconstitution, Patients will be pre-medicated as per each institution's standard protocols prior to reinfusion of PBMC products. Patient ID will be checked and verified by nursing staff and the products will be re-infused by continuous intravenous infusion pump. Patient vital signs will be monitored every 15 minutes for the duration of the procedure as per standard reinfusion protocol.
Other: ASCT — Autologous peripheral blood stem cell transplantation. (stem cells from the patient's own marrow are "harvested," stored and then returned to the body (engrafted). To be done as part of standard of care.
  Other Names: auto-SCT consolidation therapy

SUMMARY:
The purpose of this study is to explore the combination of Elotuzumab in combination with autologous stem cell transplantation and lenalidomide maintenance to see what side effects it may have and how well it works for the treatment of symptomatic multiple myeloma diagnosed and treated with induction therapy in the past year.

Induction therapy is the first phase of treatment for multiple myeloma. The goal of induction therapy for multiple myeloma is to reduce the number of plasma cells in the bone marrow and the proteins that the plasma cells produce. Induction therapy is usually given for 3-4 weeks.

An autologous peripheral blood stem cell transplant is a procedure in which immature "stem cells" are collected and stored for future use. A high dose of chemotherapy is given to the patient to destroy myeloma cells, and the patient's stem cells are replaced.

The investigational drug in this program is elotuzumab. Elotuzumab is known as BMS-901608. Elotuzumab is a manufactured protein directed against a target found on multiple myeloma cells. Lenalidomide is currently approved for patients with multiple myeloma. Melphalan and cyclophosphamide, the drugs used during stem cell collection and transplant, are also approved by the U.S. FDA. Melphalan is an FDA-approved chemotherapy for multiple myeloma and is used as high-dose treatment prior to stem cell transplantation. Cyclophosphamide is an FDA-approved chemotherapy that may be used, either alone, or in combination with other drugs to treat multiple myeloma.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, trial investigating elotuzumab and autologous PBMC reconstitution with auto-SCT consolidation therapy and lenalidomide maintenance. Fifteen patients will be enrolled in this study.

This study is based on the hypothesis that the addition of Elotuzumab and autologous PBMC reconstitution to standard-of-care auto-SCT and lenalidomide maintenance will be safe and feasible. Furthermore, we hypothesize that Elotuzumab and PBMC reconstitution will target residual myeloma cells, enhance NK cell activation and ADCC, and promote tumor-specific humoral and cellular immune responses against myeloma cells, resulting in long-term maintenance of the minimal residual disease state.

ELIGIBILITY:
Inclusion Criteria:

* Subject is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Subject has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.

Target Population

* Subjects with symptomatic MM by IMWG criteria who are receiving or have completed induction chemotherapy, who have achieved at least a PR on most recent therapy by IMWG criteria, and are eligible for auto-SCT for consolidation. A specific induction regimen is not dictated for this protocol, however, the induction regimen must not have contained melphalan (L-PAM, Alkeran).
* Age > 18 years or legal age of consent per local regulations.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2.
* Documented evidence of newly diagnosed, symptomatic MM, by IMWG criteria within one year of enrollment
* Prior lenalidomide exposure is permitted only if the subject did not discontinue lenalidomide due to a related, grade ≥ 3 AE. Age and Reproductive Status
* Men and women of childbearing potential (WOCBP) must be using 2 reliable methods of contraception to avoid pregnancy throughout the study for a period of at least 30 days before and 90 days after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. See Section 4.3.3 for the definition of WOCBP and also refer to the Revlimid Risk Management Plan guidelines.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG). The first should be performed within 10 to 14 days and the second within 24 hours prior to the start of the study drug. A prescription for lenalidomide for a female of childbearing potential must not be issued by the prescriber until negative pregnancy tests have been verified by the prescriber.
* Women must not be breastfeeding.
* Men must agree to use a latex condom and a second form of birth control during sexual contact with WOCBP, even if they have had a successful vasectomy, and must agree not to donate sperm during study drug therapy and for 90 days after therapy.
* Subjects must be willing to refrain from blood donations during study drug therapy and for 8 weeks after therapy.

Exclusion Criteria:

Target Disease

* MGUS, Waldenström's macroglobulinemia, or asymptomatic (smoldering) myeloma.
* Active plasma cell leukemia (defined as either 20% of peripheral white blood cells comprised of plasma/CD138+ cells or an absolute plasma cell count of 2 x 109/L).

Medical History and Concurrent Diseases

* All AEs of any prior chemotherapy, surgery, or radiotherapy not resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v.4.0) Grade ≤ 2.
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Acute renal failure due solely to readily reversible causes such as hypercalcemia, hyperuricemia, dehydration, hyperviscosity, or acute tubular necrosis from nephrotoxic drugs.
* Significant cardiac disease as determined by the investigator including:

  1. Known or suspected cardiac amyloidosis
  2. Congestive heart failure of Class III or IV of the NYHA classification
  3. Uncontrolled angina, hypertension or arrhythmia
  4. Myocardial infarction in the past 6 months
  5. Any uncontrolled or severe cardiovascular disease
* Prior cerebrovascular event with persistent neurologic deficit.
* Known HIV Infection or active hepatitis A, B or C.
* Any medical conditions that, in the investigator's opinion, would impose excessive risk to the subject.

Examples of such conditions include:

a. Any uncontrolled disease, such as pulmonary disease, infection, seizure disorder b. Any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent c. Active infection that requires parenteral anti-microbial or anti-parasitic treatment

* Prior or concurrent malignancy, except for the following:

  1. Adequately treated basal cell or squamous cell skin cancer;
  2. Or any other cancer from which the subject has been disease-free for > 5 years
* Uncontrolled diabetes (defined as Hgb A1C > 8.0%)
* Unable to tolerate thromboembolic prophylaxis including, as clinically indicated, aspirin, Coumadin (warfarin) or dose adjusted low-molecular weight heparin. Physical and Laboratory Test Findings
* Corrected serum calcium > 11.5 mg/dl within 2 weeks of enrollment.
* Absolute neutrophil count < 1000 cells/mm3. No granulocyte colony stimulating factors (G-CSF or GMCSF) allowed within 1 week of enrollment. No pegylated granulocyte colony stimulating factors are allowed within 3 weeks of treatment start.
* Platelets < 75,000 cell/mm3 (75 x 109/L). Qualifying laboratory value must occur at most recent measurement before enrollment and must be no more than 14 days before enrollment. No transfusions are allowed within 72 hours before qualifying laboratory value.
* Hemoglobin < 8 g/dL. Qualifying laboratory value must occur at most recent measurement before enrollment and must be no more than 14 days before enrollment. No transfusions are allowed within 72 hours before qualifying laboratory value.
* Total bilirubin > 2X ULN ,or direct bilirubin > 2.0 mg/dL.(except patients with Gilbert's syndrome then total bilirubin >2X ULN allowed in the absence of other hepatic signs or symptoms)
* AST or ALT > 3X ULN.
* CrCl < 60 ml/min by Cockcroft-Gault Formula Prior Therapy or Surgery
* Major surgery within 3 weeks prior to treatment.
* Kyphoplasty or vertebroplasty within 1 week of enrollment.
* Prior allogeneic stem cell transplant
* Treatment with plasmapheresis within 4 weeks before enrollment.
* Prior therapy with elotuzumab or any IMiD (including pomalidomide), except for prior thalidomide or lenalidomide (as defined in inclusion criteria).
* NSAIDs, IV contrast, aminoglycosides, or other potentially nephrotoxic drugs within 2 weeks of enrollment.
* Steroids within 3 weeks of enrollment, except:

  1. ≤ 10 mg prednisone or equivalent per day
  2. Steroid with little to no systemic absorption (ie, topical or inhaled steroids) Allergies and Adverse Drug Reaction
* Known hypersensitivity to lenalidomide, dexamethasone, any excipients in the elotuzumab formulation (sodium citrate, citric acid, sucrose and polysorbate 80) or recombinant protein.
* History of Grade 4 rash associated with thalidomide treatment. Sex and Reproductive Status
* Women of childbearing potential (WOCBP) who are pregnant or lactating or unwilling to use 2 forms of effective birth control.
* Men who are fertile and sexually active unwilling to use 2 forms of effective birth control if their partners are WOCBP. Other Exclusion Criteria
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Incidence of completion of treatment | up to 24 months
  Safety and tolerability will be measured by the number of evaluable patients who complete the treatment protocol.

SECONDARY OUTCOMES:
IFE level | up to 24 months
  Immunofixation Serum Test (IFE) level
sFLC level | up to 24 months
  Serum Free Light Chain analysis (sFLC) level
Bone marrow MRD analysis | up to 24 months
  Bone marrow disease (MRD) is the name for small numbers of leukaemic cells in the bone marrow
Progression-Free Survival | up to 24 months
  number of participants at 24 months who are progression-free
CyTOF mass cytometry | up to 24 months
  Immune cell reconstitution will be assessed by Cytometry by Time-Of-Flight (CyTOF) mass cytometry. This method quantifies and characterizes all cellular immune compartments.
SPEP level | up to 24 hours
  Serum protein electrophoresis (SPEP) level

CONTACTS AND LOCATIONS:
Overall Officials: Hearn Jay Cho, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Coffey DG, Osman K, Aleman A, Bekri S, Kats S, Dhadwal A, Catamero D, Kim-Schulze S, Gnjatic S, Chari A, Parekh S, Jagannath S, Cho HJ. Phase 1 study combining elotuzumab with autologous stem cell transplant and lenalidomide for multiple myeloma. J Immunother Cancer. 2024 Apr 12;12(4):e008110. doi: 10.1136/jitc-2023-008110. PMID 38609316